CLINICAL TRIAL: NCT01080547
Title: Randomized Controlled Trial Comparing Conventional and Fast Track Multi-Discipline Treatment Interventions for Colorectal Cancer
Brief Title: Study Comparing Conventional and Fast Track Multi-Discipline Treatment Interventions for Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Ding Ke-Feng, Professor of SAHZU, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009C13017
Record Dates: First submitted 2010-03-01; First posted 2010-03-04 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2016-12

CONDITIONS: Length of Stay; Complications; Adverse Drug Event; Quality of Life; Hospital Costs
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Laparoscopy; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Conventional Treatment （Laparoscopic） (Active Comparator): Randomized group of patients receiving laparoscopic colectomy with conventional perioperative treatment and mFolfox6 chemotherapy.
  Interventions: Procedure: Laparoscopic Surgery for Colorectal Cancer; Drug: mFolfox6 chemotherapy; Other: Conventional Perioperative Treatment
- FTMD Treatment （Laparoscopic） (Active Comparator): Randomized group of patients receiving laparoscopic colectomy with Fast Track Multi-Displine（FTMD）treatment and XELOX chemotherapy.
  Interventions: Procedure: Laparoscopic Surgery for Colorectal Cancer; Drug: XELOX Chemotherapy; Other: Fast Track Perioperative Treatment
- Conventional Treatment（Open Surgery） (Active Comparator): Randomized group of patients receiving open colectomy with conventional perioperative treatment and mFolfox6 chemotherapy.
  Interventions: Drug: mFolfox6 chemotherapy; Other: Conventional Perioperative Treatment; Procedure: Open Surgery for Colorectal Cancer
- FTMD Treatment（Open Surgery） (Active Comparator): Randomized group of patients receiving open colectomy with Fast Track Multi-Displine（FTMD） treatment and XELOX chemotherapy.
  Interventions: Drug: XELOX Chemotherapy; Other: Fast Track Perioperative Treatment; Procedure: Open Surgery for Colorectal Cancer

INTERVENTIONS:
Procedure: Laparoscopic Surgery for Colorectal Cancer — Laparoscopic surgery for colorectal cancer using STORZ laparoscope
  Other Names: STORZ laparoscope
  Arms: Conventional Treatment （Laparoscopic）; FTMD Treatment （Laparoscopic）
Drug: XELOX Chemotherapy — XELOX chemotherapy
  Other Names: Capecitabine; Oxaliplatin
  Arms: FTMD Treatment （Laparoscopic）; FTMD Treatment（Open Surgery）
Drug: mFolfox6 chemotherapy — Conventional (mFolfox6) chemotherapy
  Other Names: Oxaliplatin
  Arms: Conventional Treatment （Laparoscopic）; Conventional Treatment（Open Surgery）
Other: Fast Track Perioperative Treatment — Fast track treatment during perioperation period
  Other Names: Fast track surgery
  Arms: FTMD Treatment （Laparoscopic）; FTMD Treatment（Open Surgery）
Other: Conventional Perioperative Treatment — Conventional treatment during perioperation period
  Other Names: Traditional Perioperative Treatment
  Arms: Conventional Treatment （Laparoscopic）; Conventional Treatment（Open Surgery）
Procedure: Open Surgery for Colorectal Cancer — Open surgery for colorectal cancer using conventional methods
  Other Names: Traditional open surgery
  Arms: Conventional Treatment（Open Surgery）; FTMD Treatment（Open Surgery）

SUMMARY:
A new notion"Fast Track Multi-Discipline Treatment" for colorectal cancer is thought with several benefits such as shorter hospitalization stay and less costs. This randomized study aims to compare the differences between conventional and Fast Track Multi-Discipline Treatment for colorectal cancer in hospitalization day, complications, costs and quality of life.

DETAILED DESCRIPTION:
Laparoscopic Surgery, Fast Track Treatment and XELOX Chemotherapy have been introduced in the treatment of colorectal cancer. All of these procedures are contributed to reduce the hospitalization stay. However, the most economical mode for combination of these procedures is still unclear. This is a randomized controlled study, a new notion"Fast Track Multi-Discipline Treatment" is proposed, which is the combination of the Laparoscopic Surgery, Fast track perioperative treatment during perioperative period and XELOX Chemotherapy. The purpose of this study is to compare the Fast Track Multi-Discipline Treatment with the conventional treatment(Open Surgery with conventional treatment during perioperative period and mFolfox6 chemotherapy) for colorectal cancer on several aspects like the average hospitalization day, complications, costs and quality of life.The focus of the study will be to investigate whether the Fast Track Multi-Discipline Treatment reduces hospital stay with similar complications compared with conventional perioperative treatment. Moreover, the trial will clarify whether laparoscopic surgery is essential for Fast Track Multi-Discipline Treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pathologically confirmed colorectal cancer
2. Signed consent

Exclusion Criteria:

1. Tumor can be resected by endoscopic mucosal resection(EMR)
2. History of malignancy
3. Bowel obstruction or intestinal perforation
4. Evidence of metastasis by physical examination, chest roentgenogram and computed tomography of liver and pelvis
5. Acute diseases and acute attack of chronic diseases
6. Psychiatric history
7. Deformity of spine
8. ASA score≥Ⅳ
9. Mid-low rectal cancer
10. Pregnant woman
11. Needing to use Chinese traditional patent drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2010-03; Primary Completion 2014-04 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
hospitalization day | 6-month post surgery
  The overall hospitalization stay during treatment from the first day in hospital to leave hospital when finish adjuvant chemotherapy or surgery (for patients who don't need chemotherapy).

SECONDARY OUTCOMES:
surgical complications | 3-month post surgery
  Surgical complications include injury of ureter, intraoperative transfusion, infection of incision and anastomotic leakage etc.
chemotherapy related adverse event | 6-month post surgery
  Chemotherapy related adverse event, according to NCI CTCAE Version 3.0, include nausea, vomit, diarrhea and neutropenia etc.
quality of life | preoperation, 3-month post surgery and 6-month post surgery
  Quality of life will be measured by EORTC QLQ-C30 and QLQ-CR38 questionaire.
hospitalization costs | 6-month post surgery
  The overall hospitalization costs from the first day in hospital to day that adjuvant chemotherapy finished.

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Feng Ding, PhD/MD, Study Chair — The Second Affiliated Hospital, and The Key Laboratory of Cancer Prevention and Intervention, China National Ministry of Education, Zhejiang University College of Medicine.
Locations (2):
- China (2):
  - Second Affiliated Hospital Zhejiang University College of Medicine, Hangzhou, Zhejiang
  - People's Hospital of Shaoxing, Shaoxing, Zhejiang

REFERENCES:
- [Derived] Li J, Kong XX, Zhou JJ, Song YM, Huang XF, Li GH, Ying XJ, Dai XY, Lu M, Jiang K, Fu DL, Li XL, He JJ, Wang JW, Sun LF, Xu D, Xu JY, Chen M, Tian Y, Li JS, Yan M, Yuan Y, Ding KF. Fast-track multidisciplinary treatment versus conventional treatment for colorectal cancer: a multicenter, open-label randomized controlled study. BMC Cancer. 2019 Oct 23;19(1):988. doi: 10.1186/s12885-019-6188-x. PMID 31647032
- [Derived] Xu D, Li J, Song Y, Zhou J, Sun F, Wang J, Duan Y, Hu Y, Liu Y, Wang X, Sun L, Wu L, Ding K. Laparoscopic surgery contributes more to nutritional and immunologic recovery than fast-track care in colorectal cancer. World J Surg Oncol. 2015 Feb 4;13:18. doi: 10.1186/s12957-015-0445-5. PMID 25649903
- [Derived] Zhou JJ, Li J, Ying XJ, Song YM, Chen R, Chen G, Yan M, Ding KF. Fast track multi-discipline treatment (FTMDT trial) versus conventional treatment in colorectal cancer--the design of a prospective randomized controlled study. BMC Cancer. 2011 Nov 24;11:494. doi: 10.1186/1471-2407-11-494. PMID 22111914